CLINICAL TRIAL: NCT03827174
Title: Vocational Rehabilitation and Return to Work in Patients With Chronic Pain: a Randomised Controlled Trial
Brief Title: Return to Work in Patients With Chronic Pain
Acronym: UWORKin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All clinicial studies were stopped during the Covid-19 pandemic. Interventions not possible to perform, neither at workplace nor at the gym.
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); AFA Insurance (Industry); The Swedish Research Council (Other Government); Uppsala County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Pernilla Asenlof, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 160069 (AFA)
Record Dates: First submitted 2019-01-24; First posted 2019-02-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Pain; Endometriosis
Keywords: Chronic pain; Endometriosis; Opioid therapy; Return to work; Vocational rehabilitation; Behavioural medicine
MeSH Terms: conditions — Chronic Pain; Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The outcomes assessors are blinded to study condition during all measurements. Participants and providers of the return to work coordination intervention are blinded until a rehabilitation plan has been completed. Thereafter allocation to study condition is disclosed and the other components of the behaviour change ability programme are provided to those in the experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison intervention (Active Comparator): Return To Work Coordination: external and internal coordination regarding sick leave. Establishment of a common return to work plan between employer and employee.
  Interventions: Other: Return To Work Coordination
- Experimental intervention (Experimental): Return To Work Coordination + Behaviour Change Ability Programme
  Behaviour Change Ability Programme:
  1. Return to work coordination
  2. Education for employers and employees in pain neuroscience, validation, and problem-solving
  3. Patient specific goal setting for return to work
  4. Exercise and behavioural skills training related to return to work
  Interventions: Other: Return To Work Coordination; Behavioral: Behaviour Change Ability Program

INTERVENTIONS:
Other: Return To Work Coordination — External and internal coordination regarding sick leave. Establishment of a common return to work plan between employer och employee.
Behavioral: Behaviour Change Ability Program — 1. Return to work coordination
  2. Education for employers and employees in pain neuroscience, validation and problem-solving.
  3. Patient-specific goal setting for return to work
  4. Exercise and behavioural skills training related to return to work
  Arms: Experimental intervention

SUMMARY:
This study aims to evaluate whether a vocational behaviour change ability programme has any additional effect on return to work compared with return to work coordination only in persons with chronic pain.

DETAILED DESCRIPTION:
New vocational rehabilitation models including the workplace are urgently needed for persons with chronic pain.

Return to work coordination means external and internal coordination regarding sick leave by help of a rehabilitation coordinator from health care. The goal is to establish a common return to work plan between employer and employee as dictated by Swedish law. The hypothesis is that return to work coordination is not sufficient. Additional effects on return to work and work ability from a behaviour change ability programme aiming to enhance work ability by targeting context at the workplace, physical and psychological functioning, and behavioral skills at work are expected.

The hypothesis is tested in a randomised controlled trial. Before the start of the trial a series of 3-6 experimental single case studies will be performed to study the implementation of the interventions more thoroughly.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain with a duration for more than 3 months
* On sick-leave 25%-100% from salaried employment or studies, for at least 30 days
* Identified employer or director of studies
* Ability to understand, speak, and write Swedish

Exclusion Criteria:

* Severe substance use disorder
* Severe psychiatric illness
* Recruited participants with employers who does not consent to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Return to work | Number of days during a 12-month period from baseline to 12 months post baseline.
  Average sick leave according to the Swedish Social Insurance registry, defined as net days.
Work ability | 12 months
  Self-report. Work Ability Index (WAI). The questionnaire covers 7 dimensions:
  1. current work ability compared with lifetime best
  2. work ability in relation to the demands of the job
  3. number of diagnosed illnesses or limiting conditions
  4. estimated impairment owing to diseases/illnesses or limiting conditions
  5. amount of sick leave during the last year
  6. prognosis of work ability in 2 years' time
  7. psychological resources.
  The dimensions have different scores. A total index is computed ranging from 7 to 49, where higher scores indicate higher work ability.

SECONDARY OUTCOMES:
Work Ability | Baseline, 6 months, 24 months
  Self-report. Work Ability Index (WAI). The questionnaire covers 7 dimensions:
  1. current work ability compared with lifetime best
  2. work ability in relation to the demands of the job
  3. number of diagnosed illnesses or limiting conditions
  4. estimated impairment owing to diseases/illnesses or limiting conditions
  5. amount of sick leave during the last year
  6. prognosis of work ability in 2 years' time
  7. psychological resources
  The dimensions have different scores. A total index is computed ranging from 7 to 49, where higher scores indicate higher work ability.
Return to work | Baseline, 6 months, 24 months
  Average sick leave according to the Swedish Social Insurance registry, defined as net days.
Short-term sick leave < 2 weeks, number of days | 6 months, 12 months, 24 months
  Self-reported number of days with sick-leave not exceeding two weeks
Health-related quality of life: EQ-5D | Baseline, 6 months, 12 months, 24 months
  Self-report. The EuroQoL - Five dimension (EQ-5D). The five dimensions are: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each scales ranges from 0 to 2, where a low score indicates better health. The EQ-5D questionnaire also includes a visual analog scale where perceived health status is rated with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Opioid use | Baseline, 6 months, 12 months, 24 months
  Interview: Time-Line-Follow-Back. 4-week recall regarding opioid medication yes/no and dose.
Substance use disorder | Baseline, 6 months, 12 months, 24 months
  Interview: Mini International Neuropsychiatric Interview, Part J (Substance use). Response format yes/no.
  Mild substance use disorder = 2-3 symptoms Moderate substance use disorder = 4-5 symptoms Severe substance use disorder = 6 or more symptoms
Pain severity: The Brief Pain Inventory | Baseline, 6 months, 12 months, 24 months
  Self-report. The Brief Pain Inventory. Severity is measured with 4 items where worst, least, average, and current pain during the past week are scored. Each scale ranges from 0-10, where 0 = 'no pain' and 10 = 'pain as bad as can be'. Each of the severity scales will be presented separately.
Pain interference: The Brief Pain Inventory | Baseline, 6 months, 12 months, 24 months
  Self-report. The Brief Pain Inventory. Interference is measured with 7 items (general activity, mood, working ability, normal work, relations with other people, sleep, and enjoyment of life). Each scale ranges from 0 to 10, where 0 ='does not interfere', and 10 = 'completely interferes'. Interference is scored as the mean of the seven interference items. Higher scores indicate higher pain interference.
Balance | Baseline, 6 months, 12 months
  The MiniBESTest
Functional lifting capacity | Baseline, 6 months, 12 months
  Progressive Isoinertial Lifting Evaluation (PILE): cervical lifting test
Grip strength | Baseline, 6 months, 12 months
  Dynamometer GRIPPIT (name of brand)
Catastrophizing | Baseline, 6 months, 12 months
  Self-report, The Pain Catastrophizing Scale (PCS) - Swedish version. 13 items, ranging from 0 to 4 where 0 = 'not at all', 4 = 'all the time'. A total score is calculated ranging from 0 to 52 where higher scores indicate higher catastrophizing.
Fear of movement and reinjury | Baseline, 6 months, 12 months
  Self-report, The Tampa Scale of Kinesiophobia-11 (TSK-11), Swedish version. 11 items ranging from 1 to 4 where 1 = 'does not agree at all', 4 = 'totally agree'. A total score is calculated ranging from 11 to 44 where higher scores indicate higher fear of movement/kinesiophobia.
Psychological inflexibility in pain | Baseline, 6 months, 12 months
  Self-report. Psychological inflexibility in pain (PIPS) is a 12-item scale used to assess psychological inflexibility (i.e. avoidance, acceptance, fusion, values orientation, dirty discomfort) in people with chronic pain. Two main components are measured: 1) Avoidance of pain (items: 1,2,4,5,7,8,10,11), 2) Fusion with pain thoughts (items: 3,6,9,12) Scoring: Respondents are asked to rate items on a 7-point scale that ranges from 1= 'never true' to 7 = 'always true'. Scores are summed to a total score and to two subscale scores. Higher scores indicate greater levels of psychological inflexibility.
Depressive symptoms | Baseline, 6 months, 12 months, 24 months
  Self-report: Patient Health Questionnaire - 9 (PHQ-9), Swedish version. 9 items ranging from 0 ='not at all', to 3 ='almost every day'. 1 item ranging from 0 ='no difficulties, to 3 = 'extreme difficulties'. The first 9 items are summed to a sum score ranging from 0 to 27, where: 0-4 = no signs of depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression, 20-27 = severe depression. Item 10 is reported as a single item where high scores indicate high interference with daily function.
Generalised Anxiety Disorder | Baseline, 6 months, 12 months, 24 months
  Self-report: Generalised Anxiety Disorder (GAD-7). 7 items ranging from 0 ='not at all', to 3 ='almost every day'. 1 item ranging from 0 ='no difficulties, to 3 = 'extreme difficulties'. 1 item ranging from 0 ='not at all, to 3 = 'very disturbing'. The first 7 items are summed to a sum score ranging from 0 to 21, where: 0-4 = no signs of anxiety, 5-9 = mild GAD, 10-14 = moderate GAD, 15-21 = severe GAD. Item 8 is reported as a single item where higher score means higher interference.
Experience of injustice | Baseline, 6 months, 12 months
  Self-report: Injustice Experience Questionnaire (IEQ), Swedish version. 12 items ranging from 0 ='never, to 4 ='all the time'. A total score is computed by summing the scores to all 12 items, ranging from 0-48 where higher scores indicate higher experience of injustice.
  Two subscales is used. 1) Blame/unfairness by summing items 3, 7, 9, 10, 11, 23.
  2) Severity/irreparability by summing 1, 2, 4, 5, 6, 8.
Cognitive function | Baseline, 6 months, 12 months
  The Cambridge Neuropsychological Test Automated Battery (CANTAB): Spatial Working Memory, Paired Associates Learning, Delayed Match to Sample and Stocking of Cambridge (SOC).
Physical activity level | Baseline, 6 months, 12 months
  Accelerometer during one week. Time spent in sedentary, low, moderate and vigorous physical activity.
Sleep | Baseline, 6 months, 12 months
  Sleep pattern: Actigraph during night and days for one week.
Global goal achievement | 6 months, 12 months, 24 months
  Self-report. Patient global impression of change (PGIC). The measure reflects participant's beliefs about the efficacy of treatment. The patient rates overall improvement on a 7-point scale where 3 = 'very much improved', 2 = 'much improved', 1 = 'minimally improved', 0 = 'no change', -1 = 'minimally worse', -2 = 'much worse', and -3 ='very much worse'.
Explorative identification of change in biomarkers | Changes from baseline to 6 months.
  Biomarkers will be explored by use of the OLINK (name of brand) panel which enables analysis of 92 inflammation-related protein biomarkers.

OTHER OUTCOMES:
Patient-specific goals for return to work | Baseline, 6 months, 12 months
  Patient Goal Priority Questionnaire (PGPQ-WORK). Patient-specific questionnaire where the participant list 1-3 work-related activities that he or she wish to be able to perform better as a result of treatment. Activity, self-efficacy, fear of performance, and expected outcome level is then rated for each activity separately on 4 11-point numerical rating scales where higher scores indicate worse outcomes.
Self-efficacy to support return to work (employer): Number of items | Baseline, 6 months
  Study specific questions regarding the employer's self-efficacy to support the employee to return to work. Number of items is tied to individual process analysis of what is required to return to work in each specific case.
Number of participants who report adverse events associated with treatment | Up to 6 months
  Adverse events will be measured with a study-specific diary including a check-list and open ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Åsenlöf, Professor, Principal Investigator — Department of Neuroscience, Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request.